CLINICAL TRIAL: NCT03928561
Title: Efficacy of Air Cleaners in Asthmatics Allergic to Cat in ALYATEC Environmental Exposure Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SEB-001
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2019-04

CONDITIONS: Asthma; Allergy
Keywords: Asthma; Cat allergy; Environmental Exposure Chamber; Air cleaner
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, double-blind placebo-controlled study including 24 cat-asthmatic patients with GINA 1 asthma.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 - Active air cleaner then Placebo (Experimental): Exposure to cat allergen in the presence of active air cleaners then placebo. 3-week wash-out period between the two exposures.
  Interventions: Device: Active intense Pure Air XL air cleaner; Device: Placebo Intense Pure Air XL air cleaner
- 2 - Placebo then active air cleaner (Experimental): Exposure to cat allergen in the presence of placebo then active air cleaners. 3-week wash-out period between the two exposures.
  Interventions: Device: Active intense Pure Air XL air cleaner; Device: Placebo Intense Pure Air XL air cleaner

INTERVENTIONS:
Device: Active intense Pure Air XL air cleaner — Cat allergen is nebulized in the EEC. When the concentration is stable, air cleaners are switched on. The number of air cleaners placed in the EEC is defined according to the volume of the EEC and the air renewal. Patients are exposed to cat allergen in the presence of active air cleaners in the EEC
Device: Placebo Intense Pure Air XL air cleaner — Cat allergen is nebulized in the EEC. When the concentration is stable, placebo air cleaners are switched on. The placebo effect is obtained thanks to the removal of air cleaners filters prior to the exposure. The number of placebo air cleaners placed in the EEC is defined according to the volume of the EEC and the air renewal. Patients are exposed to cat allergen in the presence of placebo air cleaners in the EEC.

SUMMARY:
The aim of this study is to determine the efficacy of Rowenta® "Intense Pure Air XL" air cleaner on the early and late bronchial response, in cat-allergic asthmatic patients during an allergen exposure in ALYATEC environmental chamber (EEC)

DETAILED DESCRIPTION:
A monocentric, double-blind, placebo-controlled, cross-over study conducted outside of the pollen season. The study lasts 3 months for each patient, which includes a screening period, two exposure visits in the Alyatec Environmental Exposure Chamber (EEC) with active or placebo air cleaners, and a follow-up visit.

Patients with early asthmatic reaction during baseline exposure are randomly allocated to one of two sequences: active air cleaners /placebo or placebo/active air cleaners. Randomization is balanced (1:1) between the two sequences. There is a 3-week wash-out period between the two exposures.

ELIGIBILITY:
Inclusion Criteria:

* Controlled intermittent asthma (step 1 treatment, according to GINA Guideline 2016) with or without association with cat allergy related rhino-conjunctivitis;
* Sensitization to cat allergen extract as defined by skin prick test for cat extract with a wheal diameter of ≥3 mm greater than negative control (ALK, HØrsholm, Denmark) and specific IgE anti Fel d 1 ≥ 0.7 kU/L ( ImmunoCAP, Thermofisher, Uppsala, Sweden);
* FEV1 ≥ 70% of the predicted value;
* No cat exposure at home or outside of the home during the study;
* Positive methacholine challenge test performed using an AeroDoseur DTF-Atomisor ATO-AD 12 (Saint-Etienne, France);
* Early asthmatic response during baseline cat allergen exposure.

Exclusion Criteria:

* Uncontrolled asthma, asthma control test inferior to 20 within the 4 weeks preceding the study.
* Uncontrolled asthma 2 weeks after stopping LABA treatment.
* LABA treatment within the 2 weeks preceding the study.
* Severe asthma (> GINA 2)
* Subject lives with a cat
* Cat desensibilisation within the 6 previous months.
* Active smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Frequency of early asthmatic response | Week 9
  In subjects exposed in the EEC to an average cat allergen concentration of 40 ng/m3 (Feld1) in presence of an active air cleaner compared to a placebo.
  Early asthmatic response is defined by a drop of at least 20% compared to baseline FEV1.

SECONDARY OUTCOMES:
Frequency of late asthmatic response | Week 9
  Late asthmatic response is defined by a 15% drop of FEV1 compared to baseline FEV1 between 1h and 6h after the end of the allergen exposure.
Severity of early and/or late asthmatic response | Week 9
  Evaluated by the maximum percentage of drop in FEV1. It was measured in subjects exposed to cat allergen with active air cleaners compared to placebo air cleaners.
Difference of asthma symptoms during exposure to cat allergen with active air cleaners versus placebo. | Week 9
  The intensity of asthma symptoms is assessed using the visual analogue scale (VAS). The VAS is based on one question which allows to evaluate the symptoms on a scale from 0 to 10. 0 means no symptoms (best condition) and 10 means high symptoms (worse condition).
Difference of rhinitis symptoms during exposure to cat allergen with active air cleaners versus placebo. | Week 9
  The intensity of rhinitis symptoms is assessed using the TNSS (Total Nasal Symptom Score) nasal self-assessment questionnaire. The score of the TNSS varies from 0 (no symptoms) to 12 (high symptoms).
Difference of rhinitis symptoms during exposure to cat allergen with active air cleaners versus placebo. | Week 9
  The intensity of rhinitis symptoms is assessed using the visual analogue scale (VAS). The VAS is based on one question which allows to evaluate the symptoms on a scale from 0 to 10. 0 means no symptoms (best condition) and 10 means high symptoms (worse condition). A difference of 23 mm between two assessments done before and after exposure is considered as clinically significant.
Difference of conjunctivitis symptoms during exposure to cat allergen with active air cleaners versus placebo. | Week 9
  The intensity of conjunctivitis symptoms is assessed using the TOSS (Total Ocular Symptom Score) conjunctival self-assessment questionnaire. It varies between 0 (no symptoms) and 6 (high symptoms).
Difference of conjunctivitis symptoms during exposure to cat allergen with active air cleaners versus placebo. | Week 9
  The intensity of conjunctivitis symptoms is assessed using the visual analogue scale (conjunctivitis VAS). The VAS is based on one question which allows to evaluate the symptoms on a scale from 0 (no symptoms) to 10 (high symptoms).
Difference of conjunctivitis symptoms during exposure to cat allergen with active air cleaners versus placebo. | Week 9
  The intensity of conjunctivitis symptoms is assessed using Abelson's Score. Abelson's score varies from 0 (no symptoms) to 13 (higher symptoms). A positive conjunctival response is defined by Albelson's Score evaluated by physician above or equal to 5 during allergen exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, MD, Principal Investigator — Strasbourg University Hospital - Alyatec
Locations (1):
- Alyatec, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khayath N, Doyen V, Gherasim A, Radu C, Choual I, Beck N, Jacob A, Schoettel F, Vecellio L, Domis N, de Blay F. Validation of Strasbourg environmental exposure chamber (EEC) ALYATEC(R) in mite allergic subjects with asthma. J Asthma. 2020 Feb;57(2):140-148. doi: 10.1080/02770903.2018.1563902. Epub 2019 Mar 28. PMID 30919704
- [Derived] Gherasim A, Jacob A, Schoettel F, Domis N, de Blay F. Efficacy of air cleaners in asthmatics allergic to cat in ALYATEC(R) environmental exposure chamber. Clin Exp Allergy. 2020 Feb;50(2):160-169. doi: 10.1111/cea.13511. Epub 2019 Nov 6. PMID 31596983